CLINICAL TRIAL: NCT05603923
Title: Study of a PST-Trained Voice-Enabled Artificial Intelligence Counselor(SPEAC) for Adults With Emotional Distress (Phase 2)
Acronym: SPEAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Penn State University (Other); Washington University School of Medicine (Other); Stanford University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jun Ma, MD, PhD, Principal Investigator, Beth and George Vitoux Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1052; R33MH119237 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Lumen Coached Group (Active Comparator): Participants in this group will attend an Intervention Orientation session to receive the Coach Lumen tutorial, a study iPad, and a Lumen Intervention Workbook. They will complete 8 PST sessions with Coach Lumen using their study assigned iPad at home over 12 weeks. The first 4 sessions occur weekly and then the last 4 occur every other week. Participants will receive automated reminders on the day before and on the day of their scheduled session, and have the opportunity to reschedule sessions through the iPad. Participants will work with Coach Lumen to learn problem-solving skills to address current life challenges, plan activities, and complete home activities. Participants will also complete surveys before and after each PST session: a mood assessment survey before and a user experience survey after. At the end of study, Participants may be invited to provide their perspective regarding their Lumen use experience.
  Interventions: Behavioral: Lumen Coached PST Intervention.
- Group 2: Human Coached Group (Active Comparator): Participants in this group will receive a study iPad and Human-Coached Intervention Workbook and will complete the first of 8 PST sessions in person with a trained health coach. Participants' first PST session will be in person for approximately 1 hour. Participants will complete the remaining sessions remotely via Zoom (or by phone, if necessary) using their study iPad. The first 4 sessions occur weekly and then the last 4 occur every other week. Participants will receive automated reminder notifications on the day before and on the day of their scheduled session, and have the opportunity to reschedule sessions with their coach. Participants will also complete a mood assessment survey at the beginning of each PST session. Participants will work with their health coach to learn problem-solving skills to address current life challenges, plan activities, and complete home activities.
  Interventions: Behavioral: Human Coached PST Intervention.
- Group 3: Optional (Delayed) Lumen Coached Group (Placebo Comparator): Participants assigned to this group can choose to attend a Lumen Orientation session to receive training and a study iPad to complete 8 PST sessions with Coach Lumen after their follow-up assessment at 18 weeks. They will receive 8 Sunday mood assessment surveys to complete (4 every Sunday and then 4 every other Sunday).
  Interventions: Behavioral: Optional (delayed) Lumen Coached PST (Waitlist control).

INTERVENTIONS:
Behavioral: Lumen Coached PST Intervention. — Lumen Intervention Orientation. Participants in the Lumen intervention arm attend a Lumen orientation visit (60 minutes) during which they will be given a Lumen intervention tutorial and receive a study iPad, configured to limit access to only the Lumen intervention enabled on the device. Before leaving, participants are scheduled for the first PST session with Coach Lumen. At the end of each PST session, participants are prompted to schedule their next session with Coach Lumen. They receive automated reminder notifications 1 day prior to their next session, on the session day, and have the opportunity to make up missed sessions. As needed, Lumen intervention orientations can be done remotely.
  Arms: Group 1: Lumen Coached Group
Behavioral: Human Coached PST Intervention. — Participants in the human coached PST arm will serve as active treatment controls given the demonstrated efficacy of human coached PST in depression and anxiety. They will complete 8 PST sessions with a human coach; first session in-person and remaining sessions via videoconferencing (i.e., Zoom preferred; with phone calls allowed) on the same 4 weekly and then 4 biweekly schedule as that for Lumen participants. Participants will receive a study iPad to use for their PST sessions via zoom. Participants also complete the PHQ-9 and GAD-7 during each session. Participants will receive a certificate of completion.
  Arms: Group 2: Human Coached Group
Behavioral: Optional (delayed) Lumen Coached PST (Waitlist control). — Waitlist control participants will only complete assessments during the 18-week trial period. At the end of their 18-week assessment, they will have the option to complete 8 PST sessions on their assigned iPads.
  Arms: Group 3: Optional (Delayed) Lumen Coached Group

SUMMARY:
Approximately 200 Participants with mild-to-moderate, untreated depression and/or anxiety will be randomly assigned (by chance, like flipping a coin) to 1 of 3 study groups: Lumen Coached Problem-Solving Treatment (PST) (n=100), Human Coached PST (n=50), and optional (delayed) Lumen Coached PST as waitlist control (n=50) to improve emotional health. All participants will complete assessments at baseline and at 18 weeks post randomization.

Depending on the group assignment the PST program will be delivered by Lumen, a virtual voice-based coach on a study iPad, or by a human coach in person for the first session and then via videoconference or phone for the remaining 7 sessions. Participants assigned to the waitlist control group can receive the Lumen coached PST on a study iPad after completing their 18-week follow-up assessment.

Participants will receive 8 coaching sessions to learn problem-solving skills and work on unresolved problems in daily living that may be interfering with their emotional well-being and contributing to depression and anxiety symptoms.

DETAILED DESCRIPTION:
All participants will complete measurements of neural target engagement and treatment outcomes at both baseline (0 week) and 18 weeks.

Study Visit 1: This will include (1) Physical measurements such as height, weight, and blood pressure, (2) functional magnetic resonance imaging (fMRI) scan, (3) surveys of intervention-related measures, and (4) surveys of patient-reported outcomes, such as depressive and anxiety symptoms, social functioning, and health-related quality of life.

Following the successful completion of Visit 1 and all the surveys, participants will be randomly assigned (by chance, like flipping a coin) to 1 of 3 study groups, as described below.

Problem Solving Treatment (PST) Groups

Group 1: Lumen Coached Group :

Participants assigned to this group will attend an Intervention Orientation session to receive the Coach Lumen tutorial, a study iPad, and a Lumen Intervention Workbook. They will complete 8 PST sessions (4 weekly and then 4 biweekly) with Coach Lumen at home over 12 weeks.

Group 2: Human Coached Group Participants assigned to this group will receive a study iPad and Human-Coached Intervention Workbook, and will complete 8 PST sessions (4 weekly and then 4 biweekly) with a trained health coach over 12 weeks. They will complete the first session in person and then the remaining sessions via videoconference or phone.

Group 3: Optional (Delayed) Lumen Coached Group Participants assigned to this group may choose to attend a Lumen Orientation session to receive training and a study iPad to complete 8 PST sessions with Coach Lumen after completing their follow-up assessment at 18 weeks.

Regardless of the group assignment, participants will complete brief Nightly Mood Check-in surveys about their thoughts, feelings, and experiences over the day, for 7 nights, approximately every other week over 18 weeks (i.e., a total of 58 nights). These check-ins are sent via text message to their mobile phone.

Study Visit 2:

Regardless of group assignment, participants will be asked to attend a second in-person visit for data collection at 18 weeks. Like Visit 1, Visit 2 will include physical measurements, a brain scan (after a negative pregnancy urine test, if applicable), and online surveys (if not yet completed before the visit), and will last approximately 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Emotional distress defined by elevated depressive (PHQ-9 scores 10-19) and/or anxious symptoms (GAD-7 scores 10-14)
* Willing and able to provide informed eConsent and HIPAA authorization

Exclusion Criteria:

* Unable to speak, read, or understand English for informed consent
* Current pharmacotherapy or psychotherapy (individual or professionally led group therapy) for depression or anxiety (note: participants are not withdrawn post-randomization if they begin pharmacotherapy drugs or start psychotherapy during the study.)
* Suicidal ideation per PHQ-9 with active plan
* Bipolar or psychotic disorder, or current psychiatric treatment
* Weight ≥325 pounds due to brain scanner constraints, MRI contraindications, traumatic brain injuries, and tumor or any other known structural abnormality in the brain
* Severe medical condition (e.g., myocardial infarction or stroke or new cancer diagnosis in the past 6 months, end-stage organ failure, terminal illness) or residence in a long-term care facility
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past year
* Active alcohol or substance use disorder (including prescription drugs) based on the CAGE Questionnaire Adapted to Include Drugs (CAGE-AID)
* Cognitive impairment based on the Callahan 6-item screener
* Current or planned pregnancy or lactating (<6 months postpartum)
* Participation in other investigational treatment studies that would significantly affect participation in this study, raise safety concerns, and/or confound outcomes (participant may be asked to provide the informed consent of the other study for final decision on exclusion by a study psychiatrist)
* Family/household member of an already enrolled participant or of a study team member
* Plan to move out of the Chicago area during the study period
* Does not have reliable Wi-Fi Internet at home
* Unwillingness to user personal mobile device to receive study text messages
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Functional Magnetic Resonance Scan at 18 weeks | Baseline, 18 weeks
  Outcome Description Two neural targets defined a priori, specifically activation of the amygdala for nonconscious threat-related emotional reactivity and activation of the DLPFC for cognitive control will be assessed using fMRI. The right DLPFC is the primary neural target, while the left DLPFC and bilateral amygdala are secondary neural targets. In the facial emotion viewing paradigm, facial expression stimuli are standardized black and white photographs of 8 identities (4 female, 4 male) with evoked expressions of threat-related emotions (fear, anger), loss-related emotions (sadness) and reward-related emotions (happiness), along with neutral. For the Go-NoGo paradigm, the 'Go' and 'NoGo' stimuli are presented for 500 ms each with an inter-stimulus interval of 750 ms. The 2 paradigms are empirically validated probes of emotional reactivity and cognitive control, respectively.

SECONDARY OUTCOMES:
Change from Baseline Hospital Anxiety and Depression Scale (HADS) at 18 weeks | Baseline, 18 weeks
  HADS, including 7 questions for anxiety and 7 questions for depression, measures self-reported anxiety and depression in a general medical population of patients. Each item on the questionnaire is scored from 0-3 and the score for either anxiety or depression ranges between 0 and 21 with the following categories: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Total score for the entire scale (emotional distress) ranges from 0 to 42, with higher score indicating more distress.
Change from Baseline Penn State Worry Questionnaire (PSWQ) at 18 weeks | Baseline, 18 weeks
  PSWQ is a self-reported, 16-item, Likert-type scale that measures the trait of worry.
Change from Baseline Positive and Negative Affect Schedule (PANAS) at 18 weeks | Baseline, 18 weeks
  PANAS consists of two 10-item self-reported scales to measure positive and negative affect. Each item asks about the extent one has felt a positive or negative feeling on a 5-point scale of 1 (not at all) to 5 (very much).
Change from Baseline Social Problem-Solving Inventory-Revised: Short Form (SPSI-R:S) at 18 weeks | Baseline, 18 weeks
  Participants' problem solving abilities will be assessed using the reliable and valid SPSI-R:S that contains 25 items in the following 5 subscales: positive problem orientation (PPO), negative problem orientation (NPO), rational problem solving (RPS), impulsive/careless style (ICS), and avoidance style (AS). Each item is rated on a 5-point scale ranging from "not at all true of me" (0) to "extremely true of me" (4). SPSI-R:S is a short version of the long SPSI-R:L form.
Change from Baseline Dysfunctional Attitudes Scale (DAS) at 18 weeks | Baseline, 18 weeks
  DAS (Form A) is a 40-item self-reported scale that measures the presence and intensity of dysfunctional attitudes. Each item is rated a 7-point Likert scale (7 = fully agree; 1 = fully disagree). The higher the sum of the 40-items, the more dysfunctional attitudes an individual possesses.
Change from Baseline Sheehan Disability Scale at 18 weeks | Baseline, 18 weeks
  The Sheehan Disability Scale is a validated questionnaire that measures functional disability and is sensitive to treatment effects in clinical trials. Patients rate the extent to which their symptoms impair work/school, social, and family life on a visual analog scale from 0 to 10 and answer the number of days when their symptoms cause them to miss work/school and be unproductive at work/school.
Change from Baseline Work productivity and activity impairment questionnaire (WPAI) at 18 weeks | Baseline, 18 weeks
  The WPAI was created as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism and daily activity impairment attributable to general health in the past 7 days.
Change from Baseline Daily Mood | Baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 18)
  Daily end-of-day assessments will be captured over a one-week period at baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 18). During active treatment in the Lumen arm and the in-person PST arm, this will occur for 3 days prior to, the day of, and for 3 days after a scheduled PST session. For waitlist controls, this will occur for 7 days starting on Sunday of each assigned week. Daily mood will be measured using 8 mood items that capture both the arousal and valence components of the circumplex model of affect.
Change from Baseline Daily Stress | Baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 18)
  Outcome Description Daily end-of-day assessments will be captured over a one-week period at baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 18). During active treatment in the Lumen arm and the in-person PST arm, this will occur for 3 days prior to, the day of, and for 3 days after a scheduled PST session. For waitlist controls, this will occur for 7 days starting on Sunday of each assigned week. Daily stress will be assessed by report of stressors on that day; when stress is reported, the nature/characteristics of the stressor and response will be assessed. The type of stress will be assessed using a list of 12 categories of social problems, followed by reporting the perceived severity of the most salient stressor that day, and the degree to which the participant has had stressor-related thoughts (e.g., intrusive thoughts). Finally, we will capture an overall perceived stress report for each day.
Change from Baseline Daily Appraisal and Coping | Baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 18)
  Daily end-of-day assessments will be captured over a one-week period at baseline and every 2 weeks (i.e., on weeks 2, 4, 6, 8, 10, 12, and 18). During active treatment in the Lumen arm and the in-person PST arm, this will occur for 3 days prior to, the day of, and for 3 days after a scheduled PST session. For waitlist controls, this will occur for 7 days starting on Sunday of each assigned week. Two components of these assessments will capture a summary of appraisal and coping processes associated with daily experiences. The appraisal items will focus on assessing "problem orientation" or the general awareness and appraisals of problems during the day. The coping items will focus on assessing "problem-solving style" or the methods of planning and coping with the most salient problem experienced during the day.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Before all PST sessions (in weeks 1, 2, 3, 4, 6, 8, 10, 12)
  PHQ-9 is a self-administered instrument for screening, diagnosing, monitoring, and measuring the severity of depression. It rates the frequency of symptoms as "0" (not at all) to "3" (nearly every day) and has been validated for use in primary care. The PHQ-9 total score ranges from 0 to 27 and is categorized as follows: None or minimal depression 0-4, Mild depression 5-9, Moderate depression 10-14, Moderately severe depression 15-19, and Severe depression 20-27.
Generalized Anxiety Disorder Scale (GAD-7) | Before all PST sessions (in weeks 1, 2, 3, 4, 6, 8, 10, 12)
  GAD-7 is a valid and reliable 7-question scale to screen for 4 anxiety disorders: Post Traumatic Stress Disorder, Panic Disorder, Generalized Anxiety Disorder, and Social Phobia. A score of ≥10 indicates a high probability of 1 or more of these disorders.
User Experience Questionnaire-Short version (UEQ-S) | After Lumen Session 1, Session 4, Session 8
  UEQ-S is a validated instrument containing 8 items from the 26 items of the original UEQ. The 8 items are grouped into 2 subscales, pragmatic and hedonic quality (4 items each). A total value reflects the overall user experience.
Adapted Working Alliance Inventory for digital coaching interventions (WAI-Tech) | After Lumen Session 1, Session 4, Session 8
  WAI-Tech was based closely on the original 36-item WAI and uses a parallel set of 36 items rated on a 7-point scale (1 = "never" to 7 = "always") to measure the level of alliance between patient and digital coach along 3 domains: Task (12 items), Bond (12 items), and Goal (12 items). The Task subscale measures how responsive the digital coach was to the patient's focus or need. The Bond subscale measures the degree of the affective bond between patient and digital coach. The Goal subscale measures the extent to which goals were important, mutual, and capable of being accomplished. The WAI-Tech yields 3 subscale scores and 1 overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Department of Medicine, Vitoux Program on Aging and Prevention, Chicago, Illinois
  - UIMC Advanced Imaging Center, Chicago, Illinois

REFERENCES:
- [Derived] Kannampallil T, Ajilore OA, Smyth JM, Barve A, Ronneberg CR, Lv N, Kumar V, Garcia C, Aborisade G, Wittels NE, Tang Z, Chinnakotla B, Xiao L, Ma J. Effect and Mechanisms of a Voice-based Coach using AI on Psychological Distress: A Phase 2 Randomized Trial. medRxiv [Preprint]. 2025 Dec 29:2025.12.22.25342792. doi: 10.64898/2025.12.22.25342792. PMID 41503467
- [Derived] Ronneberg CR, Lv N, Ajilore OA, Kannampallil T, Smyth J, Kumar V, Barve A, Garcia C, Dosala S, Wittels N, Xiao L, Aborisade G, Zhang A, Tang Z, Johnson J, Ma J. Study of a PST-trained voice-enabled artificial intelligence counselor for adults with emotional distress (SPEAC-2): Design and methods. Contemp Clin Trials. 2024 Jul;142:107574. doi: 10.1016/j.cct.2024.107574. Epub 2024 May 18. PMID 38763307